CLINICAL TRIAL: NCT00736580
Title: Glove Perforation When Using Blunt vs. Sharp Needles in Cesarean Delivery
Brief Title: Glove Perforation When Using Blunt Verses Sharp Needles in Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Michael Stitely, Adjunct Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-20783
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2012-12

CONDITIONS: Cesarean Delivery; Glove Perforation
Keywords: Cesarean delivery; Surgical Needles; blunt-tip needles; surgical glove perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blunt Needles (Active Comparator): Cesarean Delivery Performed with Blunt-tipped surgical Needles
  Interventions: Other: Blunt tipped needle
- Sharp Needles (Placebo Comparator): Cesarean delivery performed with sharp surgical needles.
  Interventions: Other: Sharp needles

INTERVENTIONS:
Other: Blunt tipped needle — The Cesarean delivery is performed using blunt tipped needles.
  Arms: Blunt Needles
Other: Sharp needles — The cesarean is performed using standard sharp surgical suture needles.
  Arms: Sharp Needles

SUMMARY:
This study is assessing whether there is a decrease in surgical glove punctures using blunt tipped needles compared with sharp needles for suturing during Cesarean Delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age undergoing Cesarean Delivery

Exclusion Criteria:

* Patient less than 18 years of age.
* Patient not undergoing Cesarean Delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Stitely, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Stitely ML, Close J, Ferda A, Mehra S, Malson B, Hembree W. Glove perforations with blunt versus sharp surgical needles in caesarean delivery: a randomized trial. W V Med J. 2013 Sep-Oct;109(5):32-6. PMID 24294709

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blunt Needles | Sharp Needles
Started | 117 | 123
Completed | 117 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blunt Needles | Sharp Needles | Total
Number analyzed (Participants) | 117 | 123 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 123 | 240
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 123 | 240
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 123 | 240

OUTCOME MEASURES:

1. Primary Outcome: Surgical Glove Perforation.
Description: Direct measurement of the number of glove perforations listed by surgical case.
Time Frame: 1 week
Measure: Number; unit: Cases with a glove puncture
Arm/Group | Blunt Needles | Sharp Needles
Number analyzed (Participants) | 117 | 123
Cases with a glove puncture | 30 | 30

2. Secondary Outcome: Surgeon Satisfaction by Likert Scale.
Time Frame: 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Blunt Needles | Sharp Needles
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/123
Other Adverse Events (participants affected / at risk) | 0/117 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No